CLINICAL TRIAL: NCT01381705
Title: Validating the Predictive Value (of Response to Rituximab Induction and Maintenance) of the FCGR3A 158V/F Polymorphism Using Complimentary Genotyping Methods
Brief Title: Biomarkers in Predicting Response to Rituximab Treatment in Samples From Patients With Indolent Follicular Lymphoma
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000701978; ECOG-E4402T2
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Biological: rituximab
Genetic: DNA analysis
Genetic: gene expression analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is studying biomarkers in predicting response to rituximab treatment in samples from patients with indolent follicular lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Genotype the full cohort of samples available from the RESORT clinical trial (ECOG-E4402) for FCGR3A 158V/F in parallel to independently verify results.
* Correlate the FCGR3A 158V/F polymorphisms to response, response duration, and time to rituximab resistance.

Secondary

* Quantify copy number variation in FCGR3A in this cohort.

OUTLINE: Archived DNA samples isolate from peripheral blood mononuclear cells and from formalin-fixed paraffin-embedded tissue samples are analyzed for FCGR3A 158V/F polymorphisms using different complementary genotyping methods. Assay results are reviewed and compared with patients' outcome data.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with indolent follicular lymphoma
* Treated on RESORT trial (ECOG-E4402) comprising rituximab monotherapy and then randomized to rituximab maintenance therapy or retreatment with rituximab upon disease relapse

  * Blood and tissue samples from patients available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled in E4402 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2012-07-06 (Actual); Study Completion 2012-07-06 (Actual)

PRIMARY OUTCOMES:
Correlation of FCGR3A 158V/F polymorphisms with response, duration of response, and time to rituximab resistance | 1 year

SECONDARY OUTCOMES:
Copy number variation in FCGR3A cohort | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brad S. Kahl, MD, Principal Investigator — University of Wisconsin, Madison